CLINICAL TRIAL: NCT05989594
Title: A Home-based Mobile Guided Exercise-based Cardiac Rehabilitation Among Patients Undergoing Transcatheter Aortic Valve Replacement (REHAB-TAVR): a Randomized Clinical Trial
Brief Title: Home-based Mobile Guided Exercise-based Cardiac Rehabilitation Among Patients Undergoing TAVR
Acronym: REHAB-TAVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2022-062R
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The REHAB-TAVR group (Active Comparator): For the REHAB-TAVR group, discharge preparation will involve an exercise endurance test, exercise prescription guidance, motivational interviews, instruction on telerehabilitation, and the provision of family and peer support. Following discharge, patients will be required to adhere to their personalized exercise prescription and attend scheduled onsite follow-ups after discharge. The management model employed for this group is called home-based mobile guided exercise-based cardiac rehabilitation.
  Interventions: Behavioral: Home-based mobile guided exercise-based cardiac rehabilitation
- The Routine-TAVR group (Other): Preparation for discharge will only involve an exercise endurance test and the guidance of an exercise prescription for the Routine-TAVR group. Following discharge, nurses will conduct monthly telephone follow-ups to check on the patient's progress. Additionally, patients will be scheduled for onsite follow-ups at the Outpatient Department.
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Home-based mobile guided exercise-based cardiac rehabilitation — Discharge preparation, telerehabilitation, scheduled onsite follow-ups, telephone follow-ups, self-reporting, health education, online communication, family and peer support, mailing letters, institutional referrals, and security management.
  Arms: The REHAB-TAVR group
Behavioral: Routine Care — Discharge preparation, scheduled onsite follow-ups, telephone follow-ups
  Arms: The Routine-TAVR group

SUMMARY:
A two-parallel, evaluator-blind, single-center, randomized controlled trial was designed to assess the effectiveness of a home-based mobile guided exercise-based cardiac rehabilitation among patients undergoing Transcatheter Aortic Valve Replacement.

DETAILED DESCRIPTION:
The purpose of our study was to investigate the effect of home-based mobile-guided exercise-based cardiac rehabilitation on the improvement of exercise capacity among patients undergoing transcatheter aortic valve replacement. 90 subjects will be recruited and followed up for a six-minute walk distance, short physical performance battery, exercise adherence, quality of life, frailty, nutritional status, sleep status, readmission rate, and all-cause mortality et al. The subjects will be invited to participate in on-site visits at 1, 3, and 6 months. Patients in the interventional group will receive a home-based mobile-guided exercise-based cardiac rehabilitation for 3 months. The home-based mobile-guided exercise-based cardiac rehabilitation is a multi-component intervention strategy including the preparation for discharge, family support, motivational interviews, health education, telephone follow-up, wearable devices, APP, et al. While the patients in the control group will receive routine care. For example, the preparation for discharge of the control group does not include the guidance of mobile-guided exercise-based cardiac rehabilitation, family support, and motivational interviews. After discharge, nurses will conduct telephone follow-ups once a month for the control group. Baseline data and outcomes will be collected in a Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years and ≤ 89 years old;
* Patients scheduled to be discharged after TAVR;
* Those who have the ability to read and write, and have normal speech and communication skills;
* Patients and their families are willing to participate in this study;
* Patients or family members have the ability to use mobile and an app.

Exclusion Criteria:

* Serious complications occur before discharge (such as major bleeding, stroke, valve detachment, moderate or above perivalve leakage, coronary artery occlusion, etc.) ;
* Patients who are unable to participate in postoperative exercise rehabilitation due to limb dysfunction;
* Being in palliative care or treatment;
* Those with other Contraindication to exercise-based cardiac rehabilitation (such as resting ECG changes indicating significant ischemia, acute myocardial infarction or other acute cardiac events, unstable angina, uncontrolled arrhythmia, heart failure decompensation, etc.);
* Currently participating in other rehabilitation projects.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute Walk Distance | Month 3
  Distance walked in 6 minutes

SECONDARY OUTCOMES:
Change in 6-minute Walk Distance | Month 6
  Distance walked in 6 minutes
Change in Short Physical Performance Battery (SPPB) | Month 3 and Month 6
  The Short Physical Performance Battery is scored on a scale of 0-12, with a higher score indicating better physical function.
Exercise Adherence Assessed by the Exercise Adherence Rating Scale (EARS) | Month1, Month 3 and Month 6
  Evaluated by the Exercise Adherence Rating Scale (EARS)

OTHER OUTCOMES:
All-cause Rehospitalizations and death | Month 3 and Month 6
  The combined number of all-cause rehospitalizations and death 3 and 6 months after discharge.
Handgrip Strength | Month 3 and Month 6
  Handgrip strength is measured in kilograms by a handgrip dynamometer.
Frailty Status Assessed by the Fried Frailty Criteria | Month 3 and Month 6
  The Fried criteria consists of 5 components: low physical activity, exhaustion, weakness, slowness, and unintentional weight loss. The presence of 3 or more Fried criteria indicates frailty, 1-2 criteria indicates pre-frailty, and 0 criteria indicates no frailty.
Frailty Status Assessed by the Essential Frailty Toolset | Month 3 and Month 6
  The EFT is scored 0 (least frail) to 5 (most frail) based on the following 4 items: pre-procedural anemia, hypoalbuminemia, lower-extremity muscle weakness defined as a time of >15 s or inability to complete five sit-to-stand repetitions without using arms. and cognitive impairment is defined as a score of <24 on the Mini-Mental State Examination (which is highly unlikely if the patient is able to correctly recall 3 out of 3 words after a distractive task and may obviate the need for further cognitive testing).
Cognitive Function Assessed by the Mini-mental State Examination | Month 3 and Month 6
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding, and memory).
Quality of Life Assessed by the EuroQol 5-dimension 5-level (EQ-5D-5L) | Month 3 and Month 6
  The EQ-5D-5L is a quality-of-life tool with 5 components designed to detect health utilities: mobility, usual activities, self-care, pain/discomfort, and anxiety/depression. All components are rated on a scale of 1-5 with higher scores indicating worse health status.
Nutrition Status Assessed by the Mini-Nutritional Assessment | Month 3 and Month 6
  The Mini Nutritional Assessment (MNA) has recently been designed and validated to provide a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. The MNA test is composed of simple measurements and brief questions that can be completed in about 10 min. The sum of the MNA score distinguishes between elderly patients with 1) adequate nutritional status, MNA > or = 24; 2) protein-calorie malnutrition, MNA < 17; 3) at risk of malnutrition, MNA between 17 and 23.5.
Anxiety Assessed by the General Anxiety Disorder-7 （GAD-7） | Month 3 and Month 6
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day".
Depression Assessed by the Geriatric Depression Scale (GDS-15) | Month 3 and Month 6
  The 15-item geriatric depression scale (GDS-15) is a short form of GDS and is used to screen, diagnose, and evaluate depression in elderly individuals.
Sleep Assessed by the Pittsburgh Sleep Quality Index | Month 3 and Month 6
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.
Functional capacity Assessed by the Duke Activity Status Index (DASI) | Month 3 and Month 6
  The Duke Activity Status Index is a patient-reported estimate of functional capacity, maximal oxygen consumption (VO2 max), and maximum metabolic equivalent of tasks (METs).
Economic Analysis Assessed by direct medical costs, direct non-medical costs, and the cost of rehabilitation therapy. | Month 3 and Month 6
  Assess the economic impact of the intervention by comparing medical costs between two groups, inclusive of direct medical costs, direct non-medical costs, and the cost of rehabilitation therapy, relative to its associated changes in health outcomes.
Body Mass Index (BMI)：weight and height will be combined to report BMI in kg/m^2 | Month 3 and Month 6
  Calculate BMI values by measuring the patient's height and weight. Weight should be in kilograms. Height should be in meters)
Systolic and Diastolic Blood Pressure Assessed by a medical electronic sphygmomanometer at the outpatient. | Month 3 and Month 6
  The unit of systolic and diastolic blood pressure should be 'mmHg'.
Heart Rate Calculated by the number of heartbeats per minute. | Month 3 and Month 6
  The data collector will measure the heart rate of the patient during each outpatient visit.
New York Heart Association classification (NYHA) Presented by LevelⅠ, LevelⅡ, Level Ⅲ, Level Ⅳ. | Month 3 and Month 6
  Data collectors obtain NYHA classification by reviewing medical records.
Symptoms and Signs Assessed by the patients' self-reported whether they have palpitations, chest tightness, chest pain, dyspnea, edema, fatigue, loss of appetite, or other symptoms and signs that need to be elaborated on in detail. | Month 3 and Month 6
  During the outpatient follow-up, the patient needs to report whether they have had the symptoms and signs in the past week: yes or no. If there are other symptoms, the patient needs to write them down in detail.
Left Ventricular Ejection Fraction Assessed by the echocardiogram and presented by the unit of percentage (%) | Month 3 and Month 6
  Data collectors obtain Left Ventricular Ejection Fraction (%) by reviewing medical records.
Biomarkers for the cardiac function Assessed by N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) and Cardiac Troponin T (cTnT) | Month 3 and Month 6
  Data collectors obtain NT-proBNP and cTnT by reviewing medical records. The unit of NT-proBNP is 'pg/mL'. The unit of cTnT is 'ug/L'.
Biomarkers for renal function Assessed by Estimated Glomerular Filtration Rate (eGFR). | Month 3 and Month 6
  Data collectors obtain eGFR by reviewing medical records. The unit of eGFR is 'ml/min'.
Biomarkers for serum lipid levels Assessed by Triglyceride (TG), Cholesterol (CHOL), Low-Density Lipoprotein Cholesterol (LDL-C), and High-Density Lipoprotein Cholesterol (HDL-C). | Month 3 and Month 6
  Data collectors obtain TG, CHOL, LDL-C, and HDL-C by reviewing medical records. The unit of these biomarkers is 'mmol/L'.
Red Blood Cells (RBC) | Month 3 and Month 6
  Data collectors obtain RBC by reviewing medical records. The unit of RBC is '10^12/L'.
Haemoglobin (HGB) | Month 3 and Month 6
  Data collectors obtain HGB by reviewing medical records. The unit of HGB is 'g/L'.
White Blood Cells (WBC) | Month 3 and Month 6
  Data collectors obtain WBC by reviewing medical records. The unit of WBC is '10^9/L'.
Blood platelets (PLT) | Month 3 and Month 6
  Data collectors obtain PLT by reviewing medical records. The unit of PLT is '10^9/L'.
Biomarkers for coagulation function Assessed by Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT). | Month 3 and Month 6
  Data collectors obtain PT and APTT by reviewing medical records. The unit of PT and APTT is 's'.
Social support Assessed by the Lubben Social Network Scale-6 (LSNS-6) | Month 3 and Month 6
  The Lubben Social Network Scale-6 (LSNS-6) is a six-item, self-reported scale to assess social isolation in older adults by measuring perceived social support received by family and friends.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyun Shen, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newman-Beinart NA, Norton S, Dowling D, Gavriloff D, Vari C, Weinman JA, Godfrey EL. The development and initial psychometric evaluation of a measure assessing adherence to prescribed exercise: the Exercise Adherence Rating Scale (EARS). Physiotherapy. 2017 Jun;103(2):180-185. doi: 10.1016/j.physio.2016.11.001. Epub 2016 Nov 9. PMID 27913064
- [Result] Nagatomi Y, Ide T, Higuchi T, Nezu T, Fujino T, Tohyama T, Nagata T, Higo T, Hashimoto T, Matsushima S, Shinohara K, Yokoyama T, Eguchi A, Ogusu A, Ikeda M, Ishikawa Y, Yamashita F, Kinugawa S, Tsutsui H. Home-based cardiac rehabilitation using information and communication technology for heart failure patients with frailty. ESC Heart Fail. 2022 Aug;9(4):2407-2418. doi: 10.1002/ehf2.13934. Epub 2022 May 9. PMID 35534907
- [Derived] Shen Z, Mi S, Huang C, Zhou D, Pan W, Xu X, Lin Y, Zhang Y. Home-based mobile-guided exercise-based cardiac rehabilitation among patients undergoing transcatheter aortic valve replacement (REHAB-TAVR): protocol for a randomised clinical trial. BMJ Open. 2024 Mar 7;14(3):e080042. doi: 10.1136/bmjopen-2023-080042. PMID 38453208